CLINICAL TRIAL: NCT03529006
Title: Absorb Bioresorbable Scaffold vs. Drug Coated Balloon for Treatment Of In-Stent-Restenosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Luzerner Kantonsspital (Other)
Responsible Party: Principal Investigator, Wojciech Zasada, Clinical Trial Administrator, Luzerner Kantonsspital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AbsorbISR
Record Dates: First submitted 2018-04-19; First posted 2018-05-18 (Actual); Last update posted 2018-05-18 (Actual); Status verified 2018-05

CONDITIONS: In-stent Restenosis
Keywords: bioresorbable vascular scaffold; drug eluting balloon

ARMS (2):
- Sequent Please Drug Coated Balloon Group (Active Comparator): For Sequent Please Group, PCI (percutaneous coronary intervention) PCI procedure with Sequent Please inflation will be performed - drug eluting balloon will be used in the narrowed part of the artery. This method of treatment is one of the standard ones, which is typically used for treatment patients with diagnosis of in stent restenosis, the exact intervention and anesthesia procedures will be performed according to physician's usual practice. For bailout situation Xience stent implantation is possible.
  Interventions: Procedure: Sequent Please inflation
- Absorb Stent Group (Active Comparator): Absorb scaffold group will be treated by PCI procedure with Absorb BVS implantation - implantation of bioresorbable vascular scaffold (Absorb). Coronary stent implantation for treatment in stent restenosis is one of the standard method of treatment this disease, but Absorb system has not been investigated in this indication yet.
  Interventions: Procedure: Absorb BVS implantation

INTERVENTIONS:
Procedure: Sequent Please inflation — PCI procedure for treatment of ISR with DEB - Sequent Please - inflation
  Arms: Sequent Please Drug Coated Balloon Group
Procedure: Absorb BVS implantation — PCI procedure for treatment of ISR with Absorb BVS implantation
  Arms: Absorb Stent Group

SUMMARY:
The primary objective of this study is to demonstrate superiority of the Absorb scaffold compared to the Sequent Please Drug Coated Balloon when treating patients with In-Stent-Restenosis (ISR).

DETAILED DESCRIPTION:
Absorb ISR is randomized-controlled trial of Absorb scaffold vs. Sequent Please drug coated balloon in an all-comers population with in-stent-restenosis. The patients will be randomized in a 1:1 fashion and the investigators intend to include 150 patients.

Repeat coronary angiography will be performed 9 months post intervention in all subjects. Optical coherence tomography will be performed at baseline and at 9 months in both groups.

All patients presenting with ISR and requiring percutaneous coronary intervention will be eligible to be included in this study. This will include patients with stable angina and those presenting with acute coronary syndrome (ACS).

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Male or Female, aged 18 years or above.
* Diagnosed with ISR requiring percutaneous coronary intervention: visual diameter stenosis > 70 % and/or Fractional Flow Reserve < 0.81 and/or non-invasive testing demonstrating ischemia. This real-life population with in-stent restenosis beside typical stable patients with ISR includes ACS patients with thrombus containing lesions, patients with multivessel disease, patients with ISR in non-infarct related artery, with ISR in BMS (bare metal stent), DES (drug eluting stent) or BVS, ISR in lesion previously treated by POBA (plain old balloon angioplasty), DEB or additional stent implantation.
* Double anti-platelet therapy for the duration of at least 12 months is considered possible at the time of intervention.

Exclusion Criteria:

* Difficulty with deliver and implant the Absorb scaffold (e.g. highly calcified lesions).
* Patients who have any contraindications for using DEB (SeQent Please) or BVS (Absorb).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2015-03; Primary Completion 2016-09 (Actual); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Angiographic late lumen loss at 9 months | 9 months
  Late lumen loss will be calculated based on index and control coronary angiography.

SECONDARY OUTCOMES:
- Incidence of periprocedural complications: unplanned use of GP IIb/IIIa (Glycoprotein IIb/IIIa) inhibitors, vessel rupture, side branch occlusion, peri-procedural myocardial infarction | 9 months
  Periprocedural complications will be analyzed as combined endpoint and separately for all defined complication.
- Comparison of rate of restenosis between both groups and in specific populations (patients with acute coronary syndromes, patients with diabetes, patients with long lesions (> 25 mm)) | 9 months
  The angiographic parameter will be compared separately in all defined subgroups.
- Comparison of minimal luminal diameter between both groups and in specific populations (patients with acute coronary syndromes, patients with diabetes, patients with long lesions (> 25 mm)) | 9 months
  The angiographic parameter will be compared separately in all defined subgroups.
- Comparison of diameter stenosis between both groups and in specific populations (patients with acute coronary syndromes, patients with diabetes, patients with long lesions (> 25 mm)) | 9 months
  The angiographic parameter will be compared separately in all defined subgroups.
- Incidence of in-stent-restenosis, target lesion failure, target vessel revascularisation, stent thrombosis in in-hospital and long-term observation | 9 months
  Four clinical complications will be compared separately between study groups.
- Early, late and very late probable or definite stent thrombosis | 9 months
  Detailed description of all events of stent thrombosis will be presented.
- Cardiac and non-cardiac death in both groups | 9 months
  The frequency of deaths in both study group will be presented with differentiation according to the primary cause of the event.
- Assessment of possibility vessel measurement and stent diameter/length choice based on this measurement performed in OCT (Optical Coherence Tomography) | During index procedure.
  The usefulness of OCT for stent choice will be analyzed. The frequency of procedures, when stent choice was done based on OCT measurements will be presented.
- Result of index procedure assessment in OCT post procedure - lumen area. | During index procedure.
  The OCT parameter describing of stent implantation result during index procedure will be compared between study groups.
- Result of index procedure assessment in OCT post procedure - stent area. | During index procedure.
  The OCT parameter describing of stent implantation result during index procedure will be compared between study groups.
- Result of index procedure assessment in OCT post procedure - struts apposition assessment. | During index procedure.
  The OCT parameter - frequency of strut malapposition - describing of stent implantation result during index procedure will be compared between study groups.
- Result of index procedure assessment in OCT post procedure - dissections. | During index procedure.
  The OCT parameter describing of stent implantation result during index procedure will be compared between study groups.
- Result of index procedure assessment in OCT post procedure - stent expansion index. | During index procedure.
  The OCT parameter describing of stent implantation result during index procedure will be compared between study groups.
- OCT assessment of long-term study results - lumen area. | 9 months
  The OCT parameter describing of stent implantation result in long term FU (follow-up) will be compared between study groups.
- OCT assessment of long-term study results - stent area. | 9 months
  The OCT parameter describing of stent implantation result in long term FU (follow-up) will be compared between study groups.
- OCT assessment of long-term study results - struts apposition assessment. | 9 months
  The OCT parameter describing of stent implantation result in long term FU (follow-up) will be compared between study groups.
- OCT assessment of long-term study results - neointimal volume. | 9 months
  The OCT parameter describing of stent implantation result in long term FU (follow-up) will be compared between study groups.
- OCT assessment of long-term study results - lumen volume. | 9 months
  The OCT parameter describing of stent implantation result in long term FU (follow-up) will be compared between study groups.
- Lumen volume change between index and 9M (nine months) FU in OCT. | 9 months
  The change of OCT parameter describing of stent implantation result will be compared between index procedure and in long term FU for both study groups.
- Minimal lumen area change between index and 9M (nine months) FU in OCT. | 9 months
  The OCT parameter describing of stent implantation result will be compared between index procedure and in long term FU for both study groups.

CONTACTS AND LOCATIONS:
Overall Officials: Florim Cuculi, Principal Investigator — Luzerner Kantonsspital